CLINICAL TRIAL: NCT00413348
Title: Effect of Probiotics on Systemic Inflammation and Insulin Resistance in Type 2 Diabetics and Healthy Controls
Brief Title: Type 2 Diabetes and the Effect of Probiotics
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Royal Veterinary and Agricultural University, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: probiotics.sa.cim.rh.dk
Record Dates: First submitted 2006-12-18; First posted 2006-12-19 (Estimated); Last update posted 2006-12-19 (Estimated); Status verified 2006-12

CONDITIONS: Type 2 Diabetes; Healthy; Endotoxemia
Keywords: Type 2 diabetes; Probiotics; Insulin-resistance; Inflammation; Hyperinsulinemic euglycemic clamp; Endotoxin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Endotoxemia; Insulin Resistance; Inflammation

INTERVENTIONS:
Drug: Lactobacillus acidophilus NCFM

SUMMARY:
Insulin-resistance in type 2 diabetes is associated with chronic inflammation. Anti-inflammatory actions might increase sensitivity to insulin. Since some probiotics have anti-inflammatory properties, ingestion of the probiotic bacteria Lactobacillus Acidophilus NCFM might increase insulin-sensitivity.

The inflammatory response to endotoxin injection and the insulin-sensitivity is examined before and after four weeks ingestion of probiotics.

DETAILED DESCRIPTION:
Numerous studies have shown an association between insulin-resistance in type 2 diabetes and chronic low-grade inflammation. Some probiotics have an anti-inflammatory properties. Ingestion of probiotics might therefore, due to this property, increase sensitivity to insulin.

In this study type 2 diabetics (N=24) and healthy control (N=24) are given the probiotic bacteria Lactobacillus Acidophilus NCFM for four weeks. The anti-inflammatory effect is examined by evaluating the inflammatory response (White blood cell count, plasma-cytokines) to an iv injection of endotoxin (0,3 ng/kg) before and after the intervention. Also the insulin-sensitivity is measured with an hyperinsulinemic euglycemic clamp before and after L. acidophilus NCFM.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Type 2 diabetes

Exclusion Criteria:

* Heart failure
* Lung disease
* Infections in the last two weeks before endotoxin injections.
* Treatment with antibiotics

Ages: 25 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48
Dates: Start 2006-11; Study Completion 2007-12

PRIMARY OUTCOMES:
Change in insulin-resistance
Change in inflammatory response to E. coli endotoxin injection

CONTACTS AND LOCATIONS:
Overall Officials: Anne Sofie Andreasen, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Center of Inflammation and metabolism 7641 and Intensive Care Unit 4131, Rigshospitalet, Copenhagen, Denmark